CLINICAL TRIAL: NCT00783536
Title: An Randomized, Open Label, Multicenter Study to Compare the Efficacy and Safety of the Combination of Etanercept and Methotrexate With DMARD Therapy in Subjects With Active Early Rheumatoid Arthritis
Brief Title: A Multicenter Study to Compare the Efficacy and Safety of the Combination of Etanercept and Methotrexate in Treatment of Rheumatoid Arthritis
Acronym: DOTAR
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Wyeth (Registry Contact: Clinical Trial Registry Specialist), Wyeth
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0881A1-102380
Record Dates: First submitted 2008-10-29; First posted 2008-10-31 (Estimated); Last update posted 2022-05-09 (Actual); Status verified 2009-06

CONDITIONS: Rheumatoid Arthritis
Keywords: An randomized, open label, multicenter study to compare the ef
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Etanercept; Methotrexate; Antirheumatic Agents

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): * Clinical and demographic information
  * Clinical and Laboratory information
  Interventions: Drug: Etanercept + Methotrexate
- 2 (Active Comparator): * Clinical and demographic information
  * Clinical and Laboratory information
  Interventions: Drug: DMARDS

INTERVENTIONS:
Drug: Etanercept + Methotrexate
  Arms: 1
Drug: DMARDS
  Arms: 2

SUMMARY:
This is a randomized, open label, active-comparator, parallel design, outpatient, multicenter study being conducted in Mexico. Subjects with early active Rheumatoid Arthritis (RA) who have not received treatment with a Disease-modifying antirheumatic drug (DMARD) in the previous 6 months will be eligible for the study. Study subjects will be randomized into one of two treatments groups and receive either etanercept + methotrexate or standard non-biologic DMARD therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subject age 18 years or older
2. Diagnosis of RA
3. Disease duration of ≥ 6 months and ≤ 2 years
4. Active disease at the time of randomization
5. Negative serum pregnancy test at screening if female of childbearing potential.
6. Women of childbearing potential participating in the study must use a medically acceptable form of contraception.
7. Sexually active male must agree to use a medically accepted form of contraception during the study. If partner is using and acceptable form of contraception, this criteria is not applicable.
8. Subject is capable of understanding and signing an informed consent form
9. Subject is able and willing to self-inject study drug or have a designee who can do so
10. Subject is able and willing to take oral medication 11. Subject is able to store injectable test article at 2° C to 8° C 12. Demonstrates a negative tuberculosis screening test determined by chest

Exculsion Criteria:

1. Subject has received any previous treatment with ETN or other tumor necrosis factor (TNF) antagonist
2. Subject has received any of the following DMARDs: methotrexate, leflunomide, hydroxychloroquine, chloroquine, cyclosporine, sulphasalazine, azathioprine, D-penicillamine, cyclophosphamide within the 6 months of screening visit by the rheumatologist
3. Subject has received any investigational drug within 3 months of screening visit by the rheumatologist
4. Subject has received any biologic agent in the past
5. Subject has received any live (attenuated) vaccines within 4 weeks of screening visit by the rheumatologist
6. Subject has received intra-articular corticosteroid injection within 4 weeks of screening visit by the rheumatologist
7. Subject has received bolus intramuscular/intravenous treatment with corticosteroids (>20 mg prednisone or equivalent) within 4 weeks of screening visit by the rheumatologist
8. Subject is taking > 10 mg/day of prednisone or equivalent within 4 weeks of screening visit by the rheumatologist
9. A history or active presence of any of the following items will prevent enrollment:

   Significant concurrent medical diseases including cancer or a history of cancer Renal disease (creatinine level > 175 ?mol/L) History of drug abuse or psychiatric disease that would interfere with the subject's ability to comply with the requirements of this protocol.

   History of alcohol abuse that would interfere with the subject's ability to comply with the requirements of this protocol.

   History of known liver cirrhosis, fibrosis, or fatty liver History of any viral hepatitis within 1 year of screening
10. Active presence of the following will also prevent enrollment Subject has a significant active infection or any underlying diseases that could predispose subjects to infections according to the investigators criteria Demonstrates liver function abnormality through clinical significant hepatic enzymes results ( twice the upper limits of normal).

    Subject has leucopoenia (white blood cells < 3500 x 106/L) Subject has thrombocytopenia (platelets < 125 x 109/L) Subject has a hemoglobin level of < 85 g/L Subject is scheduled for elective major surgery within the first year of study participation Pregnant or lactating women. Positive TB by PPD and abnormal chest ray
11. Subject has a history of confirmed blood dyscrasias12. Subject has any condition judged by the physician to cause this study to be detrimental to the subject.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-11; Primary Completion 2010-06 (Estimated); Study Completion 2010-06 (Estimated)

PRIMARY OUTCOMES:
Low disease activity | 6 months

SECONDARY OUTCOMES:
Effect of the combination therapy on physical function | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer